CLINICAL TRIAL: NCT00000867
Title: A Phase II, Randomized, Double Blind, Placebo-Controlled Trial of Memantine for AIDS Dementia Complex (ADC) as Concurrent Treatment With Antiretroviral Therapy
Brief Title: A Study to Evaluate the Use of Memantine In Combination With Anti-HIV Drugs to Treat AIDS Dementia Complex (ADC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 301; DAIDS-ES ID 10687
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: AIDS Dementia Complex; HIV Infections
Keywords: Drug Therapy, Combination; Administration, Oral; AIDS Dementia Complex; Zidovudine; Anti-HIV Agents; Memantine
MeSH Terms: conditions — AIDS Dementia Complex; HIV Infections | interventions — Memantine

INTERVENTIONS:
Drug: Memantine

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of memantine, an experimental drug, in improving AIDS dementia complex (ADC).

The symptoms of ADC can be improved with zidovudine (ZDV). However, ZDV therapy has been associated with significant toxicities, and the effectiveness of ZDV seems to decrease during the second and third years of therapy. The effectiveness of other antiretroviral drugs as treatment for ADC is not known, so it is important to explore alternative therapies.

DETAILED DESCRIPTION:
The signs and symptoms of the AIDS Dementia Complex can be alleviated by zidovudine (ZDV). However, ZDV therapy has been associated with significant toxicities, particularly bone marrow suppression. The efficacy of ZDV appears to decrease during the second and third years of therapy. It is not known whether this reflects cumulative toxicity. In addition, the efficacy of other antiretroviral agents remains uncertain. Hence, adjunctive therapy for cognitive and motor symptoms of AIDS is important.

Patients will be randomized to one of the following 2 arms:

Arm 1 receives memantine plus concurrent antiretroviral therapy; Arm 2 receives placebo plus concurrent antiretroviral therapy. The initial dose of memantine is increased each week for the next 3 weeks, unless a maximum tolerated dose is reached. Following a 16-week evaluation period there is a 4-week washout prior to re-assessment. After the washout period, all patients, including those formerly randomized to the placebo arm, are given the opportunity to receive an open-label, 12-week administration of memantine. [AS PER AMENDMENT 4/6/99: The open-label phase is extended by 48 weeks to a total of 60 weeks of therapy. Patients who did not receive the initial 12 weeks of open-label treatment are eligible still for the 48-week open-label treatment phase.]

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV positive.
* Have been diagnosed with AIDS dementia complex (ADC).
* Have an estimated IQ of at least 70 (before the onset of ADC) or the ability to read at a 6th grade level.
* Have impaired mental skills.
* Are age18 or older.

Exclusion Criteria

You will not be eligible for this study if you:

* Have a history of a neurologic disease unrelated to HIV infection.
* Have a history of chronic seizures or head injuries.
* Have a history of central nervous system infections.
* Have certain cancers.
* Have any psychiatric illness.
* Have an active AIDS-defining opportunistic infection.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 1996-12; Study Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradford Navia, Study Chair; Richard Price, Study Chair
Locations (19):
- United States (19):
  - UCLA CARE Center CRS, Los Angeles, California
  - Ucsf Aids Crs, San Francisco, California
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Queens Med. Ctr., Honolulu, Hawaii
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - The Univ. of Kentucky, Lexington A2405 CRS, Lexington, Kentucky
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Washington U CRS, St Louis, Missouri
  - Univ. of Nebraska Med. Ctr., Durham Outpatient Ctr., Omaha, Nebraska
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - Mt. Sinai Med. Ctr. (N.Y.) A1801 CRS, New York, New York
  - Mt. Sinai Med. Ctr. A0404 CRS, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Letendre S, Zheng J, Yiannoutsos C, Lopez A, Ellis R, Marquie-Beck J, Zimmerman J, Gendelman H, Navia B, and The ACTG 301 and 700 Study Teams. Chemokines Correlate with Cerebral Metabolites on Magnetic Resonance Spectroscopy: A Substudy of ACTG 301 and 700. CROI 2004. Abstract 29.
- [Result] Schifitto G, Navia BA, Yiannoutsos CT, Marra CM, Chang L, Ernst T, Jarvik JG, Miller EN, Singer EJ, Ellis RJ, Kolson DL, Simpson D, Nath A, Berger J, Shriver SL, Millar LL, Colquhoun D, Lenkinski R, Gonzalez RG, Lipton SA; Adult AIDS Clinical Trial Group (ACTG) 301; 700 Teams; HIV MRS Consortium. Memantine and HIV-associated cognitive impairment: a neuropsychological and proton magnetic resonance spectroscopy study. AIDS. 2007 Sep 12;21(14):1877-86. doi: 10.1097/QAD.0b013e32813384e8. PMID 17721095
- [Result] Zhao Y, Navia BA, Marra CM, Singer EJ, Chang L, Berger J, Ellis RJ, Kolson DL, Simpson D, Miller EN, Lipton SA, Evans SR, Schifitto G; Adult Aids Clinical Trial Group (ACTG) 301 Team. Memantine for AIDS dementia complex: open-label report of ACTG 301. HIV Clin Trials. 2010 Jan-Feb;11(1):59-67. doi: 10.1310/hct1101-59. PMID 20400412